CLINICAL TRIAL: NCT02399150
Title: Biomarkers in Acute Abdomen (BIOMAB)
Brief Title: Biomarkers in Acute Abdomen
Acronym: BIOMAB
Status: Completed | Type: Observational
Sponsor: Pitié-Salpêtrière Hospital (Other)
Collaborators: Association pour la Recherche et la Formation en Anesthésie Analgésie Réanimation (Other)
Responsible Party: Principal Investigator, Hausfater Pierre, Emergency Department, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: BIOMAB
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Acute Abdominal Pain
Keywords: acute abdomen; Pain; stress biomarker
MeSH Terms: conditions — Abdomen, Acute; Pain | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA and serum blood, saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Abdominal Pain: patients presenting to the ED with acute abdomen
  Interventions: Other: No intervention as observational study

INTERVENTIONS:
Other: No intervention as observational study

SUMMARY:
Background: In the emergency setting, acute abdominal pain is a diagnostic challenge, as pain is a subjective measure, and serious causes needing surgical intervention do not always meet the clinical picture. Biomarkers measuring the individual stress or pain level may aid in identifying surgical emergencies, but there are many influencing factors that have to be taken into account.

Objective: To evaluate defined stress biomarkers for their diagnostic and prognostic utility in measuring pain, and to evaluate potential influencing or confounding factors.

Design: Prospective observational study in 200 patients presenting to the emergency department with acute abdominal pain.

Estimated duration: May 2015 - May 2016 Location Setting: Emergency Department (ED) of the Hôpital Universitaire Pitié-Salpétrière, Paris, France.

Study population: 200 patients presenting to the ED with acute abdomen

Eligibility criteria:

* Inclusion criteria: Presentation at ED with acute abdominal pain, aged at least 18 years
* Exclusion criteria: no informed consent, pregnancy, homeless, no social assurance

Procedure:

Patients presenting to the ED with acute abdominal pain will be included after informed consent is given. Blood and saliva samples will be drawn initially and after 4 hours, and baseline data assessed. All diagnostic procedures results and diagnosis made by the treating physicians as well as initiated treatment will be recorded Final diagnosis and outcome will be assessed by 2-week-telephone interview.

Measurement of candidate biomarkers will be performed in collected material. Copeptin and SAA will be measured as potential biomarkers, as a control value, cortisol will be obtained. Other biomarkers will be in consideration, depending upon availability and financial aspects.

Safety evaluations: All recommendations outlined in the ICH Guidelines for Good Clinical Practice will be adhered to throughout this trial.

Sample size considerations: The number of patients of this pilote study is based on the estimate of 25 % or 50 of acute abdomen patients to have a surgical emergency.

Significance of the study: If a biomarker is found that safely discriminates between surgical urgency and harmless abdominal pain, this will spare radiologic exposure in often young patients and will aid in optimized allocation of health care resources.

ELIGIBILITY:
Inclusion Criteria:

* Presentation at ED with acute abdominal pain, aged at least 18 years

Exclusion Criteria:

* No informed consent, pregnancy, homeless, no social assurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting to the ED with acute abdomen
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
diagnostic value of biomarkers for discriminating between self-limiting abdominal pain and acute surgical emergency | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Hausfater, MD, Pr, Principal Investigator — Service d'Accueil des Urgences, CHU Pitié-Salpêtrière, AP-HP et Université Pierre et Marie Curie Paris 06, Paris
Locations (1):
- Service d'Accueil des Urgences, CHU Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Derived] Blum CA, Faron M, Paquet AL, Velly L, Brochet C, Tresallet C, Hausfater P. Biomarkers for Detecting Surgical Emergency in Acute Abdomen-A Prospective Observational Study. J Appl Lab Med. 2025 Nov 4;10(6):1537-1551. doi: 10.1093/jalm/jfaf137. PMID 41189107